CLINICAL TRIAL: NCT04899830
Title: Study of the Acceptability and Psychosocial Impact of Using a Telepresence Robot in the Living Space of Inpatients
Acronym: ROBOLINK-e
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association APPROCHE (Other)
Collaborators: LP3C, University of Rennes 2 (Unknown); COVEA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A02088-49
Record Dates: First submitted 2021-05-10; First posted 2021-05-25 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Motor Disorders; Cognitive Disability
MeSH Terms: conditions — Motor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Installation of a telepresence robot in the home of a disabled person hospitalized in a PRM center (Experimental): From the application installed on a tablet, the patient hospitalized in a center for a period of at least 2 months can start from the center where he is hospitalized the mobile robotic telepresence assistance device installed at home to communicate with his family, his friends, his neighbors,…)
  Interventions: Device: Telepresence robot

INTERVENTIONS:
Device: Telepresence robot — From the application installed on a tablet, the patient hospitalized in a center for a period of at least 2 months can start from the center where he is hospitalized the mobile robotic telepresence assistance device installed at home to communicate with his family, his friends, his neighbors,…)

SUMMARY:
This study focuses on the mobile robot assist device for tele-interaction: the "COVEALINK 2" robot. This telepresence robot is designed for remote use inside the home. It works with an Internet connection (Wifi or 4G). It consists of a control interface (an application installed on the smartphone or tablet of the hospitalized patient) and a mobile robot placed in the home of the hospitalized patient (composed of a mobile platform, a visualization screen whose tilt is adjustable remotely for better adaptation to the interlocutors and an audio communication system). From the app installed on his smartphone or tablet, the patient hospitalized in the center for a long time (2 months minimum) will be able to start remotely (from the center where he is hospitalized) the robot and have it move within his home to communicate with the people present at the time of use (family, friends, neighbors etc.).

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 18 years old
* Affiliation to a social security scheme or beneficiary of such a scheme
* Having signed a free informed consent in writing
* Hospitalized in PRM for a foreseeable period of at least 60 days
* Living space compatible with the movement of the robot (verified by a home visit by the center's occupational therapist) and equipped with wifi
* Cognitive and motor functions compatible with the use of the tablet or phone independently, with learning capabilities to use the robot and the completion of questionnaires and interviews remotely
* Medically stable

Exclusion Criteria:

* Subject being in a period of exclusion from another protocol
* Mood and behavior disorders not stabilized
* Insufficient command of the French language
* Protected adults (guardianship / curatorship)
* Pregnant or breastfeeding women
* Persons deprived of their liberty
* Being unable to issue their consent
* Person who has already presented a form of addiction to technologies and / or video games

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-10-24 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the medium-term acceptance of robotic tele-interaction | At 2 months
  Measured with hospitalized patients using questionnaires developed by the LP3C (Laboratory of Psychology, Cognition, Behavior, Communication)

SECONDARY OUTCOMES:
Evaluation of the a priori acceptability of robotic tele-interaction | Day 0
  Measured with hospitalized patients using questionnaires developed by the LP3C (Laboratory of Psychology, Cognition, Behavior, Communication). Measure of the a priori acceptability on Day 0. A priori acceptability corresponds to the study of representations of the user upstream of any use of the technology.
Evaluation of the short-term acceptance of robotic tele-interaction | At 1 month
  Measured with hospitalized patients using questionnaires developed by the LP3C (Laboratory of Psychology, Cognition, Behavior, Communication). Measurement of acceptance at Day 30. The acceptance phase studies the user's judgment and impressions after the user's first interactions with the system
Measure the effects of the use of the telepresence device on the patient's perception of his environment and his psycho-thymic state. | Day 0
  This assessment is done using validated measurement scale relating to depression and anxiety: HAD scale (Hospital Anxiety and Depression). The HAD scale is an instrument used to screen for anxiety and depressive disorders. It comprises 14 items graded from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score = 21 ).To screen for anxiety and depressive symptoms, the following interpretation is used for each of the scores (A and D): - 7 or less: no symptoms - 8 to 10: doubtful symptomatology - 11 and over: definite symptomatology.
Measure the effects of the use of the telepresence device on the patient's perception of his environment and his psycho-thymic state. | Day 0
  This assessment is done using validated measurement scale relating to psychological well-being: EBEP (Psychological Well-Being Scale). The Ryff scale of psychological well-being "is constructed from six key dimensions: autonomy, mastery of the environment, personal development, positive relationships, giving meaning to one's life and acceptance of life. self. It consists of 18 items sides 1 to 6, where 6 indicating strongly agree. A high total score indicates psychological well-being.
Measure the effects of the use of the telepresence device on the patient's perception of his environment and his psycho-thymic state. | Day 0
  This assessment is done using validated measurement scale relating to quality of life: questionnaire general SF-36 (Short Form 36 Healt Survey). The SF-36 questionnaire is a multidimensional questionnaire that assesses quality of life in relation to health status, regardless of causal pathology, gender, age and treatment. It assesses functioning and overall well-being using a questionnaire using 36 questions divided into 8 dimensions (physical functioning, role limitations related to physical health, physical pain, general health, vitality, functioning or social well-being, role limitations related to mental health, mental health).
Measure the effects of the use of the telepresence device on the patient's perception of his environment and his psycho-thymic state. | Day 0
  This assessment is done using validated measurement scale relating to level of social participation: LHS scale (London Handicap Scale). This scale questions everyday life by assessing mobility, physical independence, occupation (work, hobbies, vacations, etc.), social integration, perception of the outside world and economic independence.
  It takes the form of a questionnaire comprising 6 items rated from 0 to 1: - 1 = no handicap - 0 = maximum handicap.
Measure the effects of the use of the telepresence device on the patient's perception of his environment and his psycho-thymic state. | At 2 months
  This assessment is done using validated measurement scale relating to depression and anxiety: HAD scale (Hospital Anxiety and Depression). The HAD scale is an instrument used to screen for anxiety and depressive disorders. It comprises 14 items graded from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score = 21 ).To screen for anxiety and depressive symptoms, the following interpretation is used for each of the scores (A and D): - 7 or less: no symptoms - 8 to 10: doubtful symptomatology - 11 and over: definite symptomatology.
Measure the effects of the use of the telepresence device on the patient's perception of his environment and his psycho-thymic state. | At 2 months
  This assessment is done using validated measurement scale relating to psychological well-being: EBEP (Psychological Well-Being Scale). The Ryff scale of psychological well-being "is constructed from six key dimensions: autonomy, mastery of the environment, personal development, positive relationships, giving meaning to one's life and acceptance of life. self. It consists of 18 items sides 1 to 6, where 6 indicating strongly agree. A high total score indicates psychological well-being.
Measure the effects of the use of the telepresence device on the patient's perception of his environment and his psycho-thymic state. | At 2 months
  This assessment is done using validated measurement scale relating to quality of life: questionnaire general SF-36 (Short Form 36 Healt Survey). The SF-36 questionnaire is a multidimensional questionnaire that assesses quality of life in relation to health status, regardless of causal pathology, gender, age and treatment. It assesses functioning and overall well-being using a questionnaire using 36 questions divided into 8 dimensions (physical functioning, role limitations related to physical health, physical pain, general health, vitality, functioning or social well-being, role limitations related to mental health, mental health).
Measure the effects of the use of the telepresence device on the patient's perception of his environment and his psycho-thymic state. | At 2 months
  This assessment is done using validated measurement scale relating to level of social participation: LHS scale (London Handicap Scale). This scale questions everyday life by assessing mobility, physical independence, occupation (work, hobbies, vacations, etc.), social integration, perception of the outside world and economic independence.
  It takes the form of a questionnaire comprising 6 items rated from 0 to 1: - 1 = no handicap - 0 = maximum handicap.
Evaluation of the a priori acceptability of robotic tele-interaction for users, relatives and members of the multidisciplinary team | Day 0
  Measurement with categories of users around the patient and members of the multidisciplinary team, using questionnaires developed by the LP3C (Laboratory of Psychology, Cognition, Behavior, Communication). Measurement of a priori acceptability on Day 0. A priori acceptability corresponds to the study of representations of the user upstream of any use of the technology.
Evaluation of the medium-term acceptance of robotic tele-interaction for users, relatives and members of the multidisciplinary team | At 2 months
  Measurement with categories of users around the patient and members of the multidisciplinary team, using questionnaires developed by the LP3C (Laboratory of Psychology, Cognition, Behavior, Communication). Measurement of acceptance at Day 60. The acceptance phase studies the user's judgment and impressions after the user's first interactions with the system.

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud Honoré, Doctor, Principal Investigator — CMRRF de Kerpape
Locations (4):
- France (4):
  - CR Mulhouse, Mulhouse, Alsace
  - IUR Clémenceau, Strasbourg, Alsace
  - CMRRF de Kerpape, Ploemeur, Brittany Region
  - CMPR Côte d'Amour, Saint-Nazaire, Pays de la Loire Region

IPD SHARING:
Plan to Share IPD: No